CLINICAL TRIAL: NCT06523751
Title: Determining Distal Outflow Tract Function in Open Angle Glaucoma as a Predictive Test for the Success of Ab Interno Trabeculectomy
Brief Title: Trabeculopuncture as Predictive Test for the Success of Ab Interno Trabeculectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 113-21-me
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Open Angle Glaucoma; Pseudoexfoliation Glaucoma
Keywords: Ab Interno Trabeculectomy; Trabeculopuncture; Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome

STUDY DESIGN:
Intervention Model Description: Determining Distal Outflow Tract Function in Open Angle Glaucoma as a Predictive Test for the Success of Ab Interno Trabeculectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trabeculopuncture (Experimental): Individuals undergo neodymium-doped yttrium aluminum garnet (Nd:YAG) trabeculopuncture prior to ab interno trabeculectomy.
  Interventions: Diagnostic Test: Trabeculopuncture

INTERVENTIONS:
Diagnostic Test: Trabeculopuncture — Trabeculopuncture is performed with a Nd:YAG laser on the trabecular meshwork. Four punctures are created along the 180° nasal trabecular meshwork.

SUMMARY:
The purpose of this study is to perform trabeculopuncture a test to determine the distal outflow tract function to predict the success of ab interno trabeculectomy.

DETAILED DESCRIPTION:
The aim of this study is to develop a non-invasive predictive test for the function of the distal outflow tract after ab interno trabeculectomy for open angle glaucoma. We hypothesize that the ocular pressure drop and outflow change after preoperative trabeculectomy may predict the success of ab interno trabeculectomy. The results of this study should allow trabeculopuncture to be used to select the most appropriate procedure for the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* individuals ≥ 18 years of age
* clinical diagnosis of: primary open angle glaucoma, pigmentary glaucoma, or pseudoexfoliation glaucoma
* uncontrolled intraocular pressure (IOP) with maximally tolerated medical therapy
* progressive thinning of retinal nerve fiber layer assessed by Spectral domain optical coherence tomography (p < 0.05)
* progression of visual field defects
* visually significant cataract and indication to reduce IOP or glaucoma medication burden

Exclusion Criteria:

* clinical diagnosis of neovascular glaucoma, angle-closure glaucoma, uveitic glaucoma, neovascular glaucoma
* prior glaucoma surgery
* preexisting conditions affecting the episcleral venous pressure including Grave's ophthalmopathy, Sturge-Weber syndrome, Arteriovenous fistulas (carotid-cavernous fistula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
IOP | before and two hours after trabeculopuncture, one and four weeks postoperatively (after ab interno trabeculectomy), and three months postoperatively
  Intraocular pressure measured by Goldmann applanation tonometry
Outflow facility | before and two hours after trabeculopuncture, one and four weeks postoperatively (after ab interno trabeculectomy), and three months postoperatively
  Outflow facility is measured by the use of a pneumatonometer
Surgical success | at month three
  surgical success at month three is defined as 20% IOP reduction without increasing the number of glaucoma drops

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kampik, MD, PhD, Principal Investigator — Department of Ophthalmology University Hospital Würzburg
Locations (1):
- Uniklinikum Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma-Fuehring R, Dakroub M, Han H, Hillenkamp J, Loewen NA. Trabeculopuncture as a predictive test of distal outflow resistance in canal-based surgery. Sci Rep. 2022 Jun 22;12(1):10584. doi: 10.1038/s41598-022-13990-9. PMID 35732782
- [Background] Epstein DL, Melamed S, Puliafto CA, Steinert RF. Neodymium: YAG laser trabeculopuncture in open-angle glaucoma. Ophthalmology. 1985 Jul;92(7):931-7. doi: 10.1016/s0161-6420(85)33932-5. PMID 4022580
- [Background] Melamed S, Pei J, Puliafito CA, Epstein DL. Q-switched neodymium-YAG laser trabeculopuncture in monkeys. Arch Ophthalmol. 1985 Jan;103(1):129-33. doi: 10.1001/archopht.1985.01050010135037. PMID 3977666
- [Background] Del Priore LV, Robin AL, Pollack IP. Long-term follow-up of neodymium: YAG laser angle surgery for open-angle glaucoma. Ophthalmology. 1988 Feb;95(2):277-81. doi: 10.1016/s0161-6420(88)33195-7. PMID 3173993

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT06523751/Prot_SAP_000.pdf